CLINICAL TRIAL: NCT02477423
Title: A Randomized Controlled Trial Investigating if Antibiotic Use in the First 48 Hours of Life Adversely Impacts the Preterm Infant Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB15-0053
Record Dates: First submitted 2015-06-16; First posted 2015-06-22 (Estimated); Results first posted 2020-09-03 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Premature Birth of Newborn; Enterocolitis, Necrotizing
Keywords: Microbiome; Antibiotics
MeSH Terms: conditions — Premature Birth; Enterocolitis, Necrotizing | interventions — Ampicillin; Gentamicins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Randomized & Blinded - Receiving Antibiotics (Active Comparator): The infants within this arm of the study meet the inclusion criteria as being low risk. They will be randomized to receive routine ampicillin and gentamicin for the initial 48 hours of their life as a routine rule-out sepsis. Stool samples will be collected throughout hospitalization and at 18 months of life.
  Interventions: Drug: Ampicillin; Drug: Gentamicins
- Randomized & Blinded - Receiving Placebo (Placebo Comparator): The infants within this arm of the study meet the inclusion criteria as being low risk. They will be randomized to receive placebo (saline) in place of ampicillin and gentamicin for the initial 48 hours of their life as a routine rule-out sepsis. Stool samples will be collected throughout hospitalization and at 18 months of life.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ampicillin — Ampicillin will be given as routine antibiotic coverage for those in the active arm, as the standard initial antibiotic used within the neonatal unit. It may also be used for patients who are not eligible for randomization.
  Arms: Randomized & Blinded - Receiving Antibiotics
Drug: Gentamicins — Gentamicin will be given as routine antibiotic coverage for those in the active arm, as the standard initial antibiotic used within the neonatal unit. It may also be used for patients who are not eligible for randomization.
  Arms: Randomized & Blinded - Receiving Antibiotics
Drug: Placebo — Normal saline will be given as placebo for those in the placebo comparator group.
  Arms: Randomized & Blinded - Receiving Placebo

SUMMARY:
The purpose of this study is to determine whether antibiotics given immediately after birth alter the development of the developing preterm infant's microbiome, which may further alter overall clinical outcomes.

ELIGIBILITY:
Inclusion Criteria for antibiotic randomization:

1. Infant must be born between the gestational ages of 28 0/7 weeks and 34 6/7 weeks

   -AND-
2. Infant must be born at investigator's home institution.

   -AND-
3. Infant must be considered to have a low risk of infection by one of the following criteria:

   1. Delivered for maternal indications (Cesarean section or induction of labor for maternal health, including pre-eclampsia, placental abruption, history of intrauterine fetal demise (IUFD)/abruption, multiple gestation requiring preterm delivery, etc) -OR-
   2. Delivered due to preterm labor to a mother without the diagnosis of chorioamnionitis/maternal fever or prolonged rupture of membranes >18 hours

Exclusion Criteria for antibiotic randomization:

1. Signs of clinical illness within the first 3 hours of life:

   1. 5-minute Apgar <5
   2. Requiring vasoactive drugs
   3. Seizures
   4. Significant respiratory distress requiring supplemental oxygen >40%
2. Immature:Total (I:T) Ratio of >0.2 on initial complete blood count (CBC)
3. Congenital anomalies, including renal anomalies requiring serum antibiotic level monitoring

ANY infant born between the gestational ages of 28 0/7 weeks and 34 6/7 weeks who do not meet inclusion criteria, with parental consent, can participate in the stool analysis only arm of the study.

Max Age: 6 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2015-07; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago Medical Center - Comer Children's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients in the study were enrolled from The University of Chicago Comer Children's Hospital, a level IV NICU in Chicago, Illinois, as well as Northshore University HealthSystem Evanston Hospital, a level III NICU in Evanston, Illinois from 2015-2018.
Period: Overall Study
Arm/Group | Randomized & Blinded - Receiving Antibiotics | Randomized & Blinded - Receiving Placebo
Started | 12 | 15
Completed | 11 | 11
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Randomized & Blinded - Receiving Antibiotics: The infants within this arm of the study meet the inclusion criteria as being low risk. They will be randomized to receive routine ampicillin and gentamicin for the initial 48 hours of their life as a routine rule-out sepsis. Stool samples will be collected throughout hospitalization and at 18 months of life.
  Ampicillin: Ampicillin will be given as routine antibiotic coverage for those in the active arm, as the standard initial antibiotic used within the neonatal unit. It may also be used for patients who are not eligible for randomization.
  Gentamicin: Gentamicin will be given as routine antibiotic coverage for those in the active arm, as the standard initial antibiotic used within the neonatal unit. It may also be used for patients who are not eligible for randomization.
- Total: Total of all reporting groups
Arm/Group | Randomized & Blinded - Receiving Antibiotics | Randomized & Blinded - Receiving Placebo | Total
Number analyzed (Participants) | 12 | 15 | 27
Age, Customized [Mean (Full Range); unit: weeks]
  Gestational Age | 32.6 [28.1 to 34] | 31.9 [28 to 33.9] | 32.3 [28.1 to 34]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 7 | 8 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 14 | 25
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Richness of the Preterm Infant Microbiome
Description: Number of 16S rRNA gene amplicon sequence variants (i.e., proxy for prokaryote species-like groupings) detected in each sample. A higher richness means that a higher number of species of archaea and bacteria was detected in a sample.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: 16S rRNA gene amplicon sequence variants
Arm/Group | Randomized & Blinded - Receiving Antibiotics | Randomized & Blinded - Receiving Placebo
Number analyzed (Participants) | 11 | 11
16S rRNA gene amplicon sequence variants | 12.8 (5.3) | 11 (6.9)

2. Primary Outcome: Shannon Diversity of the Preterm Infant Microbiome
Description: Function of richness and evenness of 16S rRNA gene amplicon sequence variants (i.e., proxy for prokaryote species-like groupings) within each sample. A higher Shannon diversity means that a sample had a combination of a higher number of species of archaea and bacteria, and/or a more even relative abundance of those species within a sample.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Shannon diversity
Arm/Group | Randomized & Blinded - Receiving Antibiotics | Randomized & Blinded - Receiving Placebo
Number analyzed (Participants) | 11 | 11
Shannon diversity | 5 (3.6) | 3.8 (3.3)

3. Secondary Outcome: Chronic Lung Disease of Infancy (CLD)
Description: Premature infants who require > 21% FiO2 for at least 28 days and/or at 36 weeks corrected gestation
Time Frame: 4-12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized & Blinded - Receiving Antibiotics | Randomized & Blinded - Receiving Placebo
Number analyzed (Participants) | 12 | 15
Participants | 0 | 0

4. Secondary Outcome: Necrotizing Enterocolitis (NEC)
Description: Any patient showing signs/symptoms of this acute neonatal gastrointestinal disease, including abdominal distension, bloody stools, systemic illness, and radiographic changes (pneumatosis intestinalis, portal venous gas, free intraperitoneal gas).
Time Frame: 4-12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized & Blinded - Receiving Antibiotics | Randomized & Blinded - Receiving Placebo
Number analyzed (Participants) | 12 | 15
Participants | 0 | 0

5. Secondary Outcome: Retinopathy of Prematurity (ROP)
Description: Cases of ROP as diagnosed by the pediatric ophthalmologist
Time Frame: 4-12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized & Blinded - Receiving Antibiotics | Randomized & Blinded - Receiving Placebo
Number analyzed (Participants) | 12 | 15
Participants | 0 | 0

6. Secondary Outcome: Intraventricular Hemorrhage (IVH)
Description: Cases of IVH present on any head ultrasound obtained during patient's hospitalization
Time Frame: 4-12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized & Blinded - Receiving Antibiotics | Randomized & Blinded - Receiving Placebo
Number analyzed (Participants) | 12 | 15
Participants | 0 | 0

7. Secondary Outcome: Death
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized & Blinded - Receiving Antibiotics | Randomized & Blinded - Receiving Placebo
Number analyzed (Participants) | 12 | 15
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Randomized & Blinded - Receiving Antibiotics | Randomized & Blinded - Receiving Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/15
Other Adverse Events (participants affected / at risk) | 0/12 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-08-30): https://cdn.clinicaltrials.gov/large-docs/23/NCT02477423/Prot_000.pdf